CLINICAL TRIAL: NCT04024605
Title: Bioavailability of Protein and Amino Acids From Oilseeds in Healthy Volunteers
Acronym: PRODIGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: AgroParisTech (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PRODIGE
Record Dates: First submitted 2019-02-19; First posted 2019-07-18 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Protein
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sunflower (Experimental): Biscuits containing sunflower isolate intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Sunflower
- Rapeseed (Experimental): Biscuits containing rapeseed isolate intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Rapeseed
- Flaxseed (Experimental): Biscuits containing flaxseed isolate intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Flaxseed
- Lupin (Experimental): Biscuits containing lupin flour intrinsically labelled with 15N and 2H
  Interventions: Dietary Supplement: Lupin

INTERVENTIONS:
Dietary Supplement: Sunflower — Plant proteins are intrinsically enriched with 15N and 2H. There are incorporated into biscuits. The biscuits are formulated to supply 20 g of plant protein per volunteer.
  Arms: Sunflower
Dietary Supplement: Rapeseed — Plant proteins are intrinsically enriched with 15N and 2H. There are incorporated into biscuits. The biscuits are formulated to supply 20 g of plant protein per volunteer.
  Arms: Rapeseed
Dietary Supplement: Flaxseed — Plant proteins are intrinsically enriched with 15N and 2H. There are incorporated into biscuits. The biscuits are formulated to supply 20 g of plant protein per volunteer.
  Arms: Flaxseed
Dietary Supplement: Lupin — Plant proteins are intrinsically enriched with 15N and 2H. There are incorporated into biscuits. The biscuits are formulated to supply 20 g of plant protein per volunteer.
  Arms: Lupin

SUMMARY:
The study aims to determine in healthy subjects the bioavailability of protein and amino acids of 4 protein sources: sunflower, rapeseed, lupin, flax. For this purpose, the investigators will compare two methods:

1. the standard method consisting in measuring the ileal digestibility using ileal tubes
2. an alternative method that has been proposed by an Food and Agriculture Organization (FAO) expert group: the dual isotope method

DETAILED DESCRIPTION:
4 groups of healthy volunteers are recruited (males and females from 18 to 65 y old), BMI from 18 to 30.

Each group tests a protein source (20g) incorporated in a biscuit that is divided in small portions to perform a repeated meal protocol. Protein sources (sunflower, rapeseed, flaxseed or lupin) are intrinsically labeled with 15N and deuterium (2H).

The day before the meal test, the volunteers are equipped with an intestinal tube that migrates until the ileum. On the day of the experiment, the position of the intestinal tube is checked by radiography in order to verify its location at the terminal ileum. A catheter is inserted in the forearm vein for blood sampling. A saline solution containing polyethylene glycol 4000 (PEG-4000, 20 g/L), used as a non-absorbable marker of the intestinal flow, is infused into the ileum in order to calculate the flow rate of the intestinal effluents. After a basal blood and urine sampling, as well as a basal collection of ileal effluents performed for 30 min, subject ingests at t=0 the first biscuit dose. The small biscuit portions are ingested every 30 min for 4h, to achieve an isotopic plateau. Tracer doses of carbon 13 (13C) amino acids are ingested concomitantly with the biscuit doses. Non absorbable markers are added to the test meal to correct for incomplete recovery at the ileal level.

The postprandial sampling period lasts for 8 h after the meal ingestion. The intestinal content is continuously collected over ice and pooled every 30 min. Blood is sampled every 30 min for 4 h, and hourly thereafter.Total urine is collected every 2 h.

Measurements:

In the effluents, the investigators measure PEG 4000, nitrogen (N) and 15N, carbon and 13C, amino acids (AA), 15N and 13C in amino acids and the non-absorbable markers of the meal. The investigators calculate the ileal flow rate, the overall real ileal protein digestibility and the real ileal digestibility of individual amino acids.

In the plasma, the investigators measure uremia and 15N in urea, AA and protein to measure the transfer of dietary N in plasma protein pools; 15N, 2H and 13C in individual amino acids too measure the relative bioavailability of 15N/2H amino acids compared to free 13C amino acids.

In the urine, the investigators measure urea and 15N in the urea ammonia to calculate the postprandial deamination losses.

These measurements will allow to determine the protein and amino acid bioavailability from 4 different plant protein sources, using the classical method implying ileal sampling and intrinsic tracer of dietary protein (15N). Additionally, it will allow to test a less invasive procedure using multiple tracers to assess the amino acid bioavailability.

ELIGIBILITY:
Inclusion Criteria:

* 18<BMI<30
* Healthy
* Insured under the French social security system
* for women: use of birth control
* signed informed consent

Exclusion Criteria:

* Any dietary allergy
* Latex allergy
* Positive serology to HIV, hepatite C virus antibody, hepatite B virus surface antigen and core antibodies
* Gluten intolerance
* Anemia
* Abusive use of drugs or alcohol
* Hypertension, diabetes, digestive disease, hepatic or renal disease, severe cardiac disease
* Pregnancy
* High sport practicing (>7h/wk)
* Blood donation in the 3 months prior to the study
* Participation in a clinical study in the 3 months prior to the study
* No signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of ileal digestibility of plant proteins | time -30 minutes to 8 hours after the meal
  Total N and 15N will be measured by Elemental Analyzer coupled to an Isotopic Ratio Mass Spectrometer (EA-IRMS) and the percentage of dietary N reaching the terminal ileum will be then determined. This percentage will be corrected by the ileal flow rate which is estimated with measurement of PEG concentration in effluents by a turbidimetric methods. Ileal digestibility of plant proteins (i.e. N digestibility) will be calculated as 100 - corrected dietary N percentage.
Percentage of ileal digestibility of amino acids from plant proteins | time -30 minutes to 8 hours after the meal
  Amino acid concentrations will be measured by Ultra high performance liquid chromatography (UHPLC) and 15N, 2H and 13C enrichment in individual amino acids will be measured by Gas Chromatography-Combustion-Isotope Ratio Mass Spectrometry (GC-C-IRMS) in order to determine the percentage of dietary individual amino acids reaching the terminal ileum. This percentage will be corrected by the ileal flow rate which is estimated with measurement of PEG concentration in effluents by a turbidimetric methods. Ileal digestibility of plant amino acid will be calculated as 100 - corrected dietary amino acid percentage.
Percentage of net postprandial protein utilization of plant proteins | time -30 minutes to 8 hours after the meal
  Urea in plasma and urine (by enzymatic methods) will be determined and associated with 15N enrichment values (by EA IRMS) to determine the 15N transfer in plasma and urinary N pools and calculate the net postprandial protein utilization.
Postprandial plasma kinetics of dietary amino acids | time -30 minutes to 8 hours after the meal
  Amino acids in plasma will be determined by UHPLC and associated with 15N enrichment values in individual amino acids (by GC C IRMS) to determined the kinetics of amino acids from plant proteins.
Postprandial metabolism of glucose 1 | time -30 minutes to 8 hours after the meal
  Glycemia (by enzymatic methods) will be determined in plasma.
Postprandial metabolism of glucose 2 | time -30 minutes to 8 hours after the meal
  Insulinemia (by ELISA) will be determined in plasma.

SECONDARY OUTCOMES:
Validation of the dual isotope method to assess the bioavailability of individual amino acids | time -30 minutes to 8 hours after the meal
  Measurements of 15N, 2H and 13C amino acids in the plasma by GC-C-IRMS

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Derived] Tessier R, Calvez J, Airinei G, Khodorova N, Dauguet S, Galet O, Chapelais M, Tome D, Benamouzig R, Gaudichon C. Digestive and metabolic bioavailability in healthy humans of 15N-labeled rapeseed and flaxseed protein incorporated in biscuits. Am J Clin Nutr. 2023 May;117(5):896-902. doi: 10.1016/j.ajcnut.2023.02.020. Epub 2023 Feb 24. PMID 36842754
- [Derived] Tessier R, Calvez J, Airinei G, Khodorova N, Kapel R, Quinsac A, Galet O, Piedcoq J, Benamouzig R, Tome D, Gaudichon C. The True Amino Acid Digestibility of 15N-Labelled Sunflower Biscuits Determined with Ileal Balance and Dual Isotope Methods in Healthy Humans. J Nutr. 2022 Mar 3;152(3):698-706. doi: 10.1093/jn/nxab423. PMID 34910189